CLINICAL TRIAL: NCT04691661
Title: A Randomized Double-blind Placebo-controlled Multicentre Study to Assess Safety, Tolerability, Pharmacokinetics and Efficacy of Radotinib in Parkinson's Disease
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy Study of Radotinib in Parkinson's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RT51EP1902
Record Dates: First submitted 2020-12-16; First posted 2020-12-31 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — 4-methyl-N-(3-(4-methylimidazol-1-yl)-5-trifluoromethylphenyl)-3-(4-pyrazin-2-ylpyrimidin-2-ylamino)benzamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo: Dose escalation (Placebo Comparator): Forty (40) subject will be recruited and randomized into 4 dosing groups. In each dosing group, ten (10) will be randomized and 8 of 10 will receive the active product (Radotinib) and 2 subjects will receive the matching placebo orally once daily for 6 months at each escalating dose level.
  Interventions: Drug: Placebo
- Radotinib HCl: Dose escalation (Experimental): Forty (40) subject will be recruited and randomized into 4 dosing groups. In each dosing group, ten (10) will be randomized and 8 of 10 will receive the active product (Radotinib) and 2 subjects will receive the matching placebo orally once daily for 6 months at each escalating dose level.
  The inclusion of subjects in the next dose level will be decided by the sponsor in consultation with a Data Monitoring Committee (DMC).
  Interventions: Drug: Radotinib HCl 50 mg

INTERVENTIONS:
Drug: Radotinib HCl 50 mg — Enrolled subject will continue to administer Radotinib 50mg/day, 100mg/day, 150mg/day, 200mg/day, depending on the dose level once daily for 6 months.
  Other Names: Radotinib; IY5511
  Arms: Radotinib HCl: Dose escalation
Drug: Placebo — Placebo
  Arms: Placebo: Dose escalation

SUMMARY:
This is a safety, tolerability, pharmacokinetic and efficacy study in subjects with Parkinson's disease

DETAILED DESCRIPTION:
This study is will be conducting to determine if Radotinib is safe and can be tolerated by patients with Parkinson's disease (PD) and to learn if Radotinib can be potential therapeutic agents for the treatment of PD.

Radotinib has been approved by Ministry of Food & Drug Safety of Korea to treat Chronic Myeloid Leukemia (CML) but it has not been approved for PD.

In nonclinical efficacy study, therapeutic effect of Radotinib HCl, c-Abl inhibitor, which exhibits improved pharmacokinetic properties and BBB penetration compared to nilotinib and other c-Abl inhibitors, was tested in a preclinical α-synuclein preformed fibrils (PFF) model of sporadic PD. As a result, the treatment of Radotinib HCl protects the α-synuclein PFFs-induced neuronal toxicity, reduces the PFFs-induced LB/LN-like pathology, and inhibits the PFFs-induced c-Abl activation in neurons. In vivo studies demonstrate that administration of Radotinib HCl prevents dopamine neuron loss and behavioral deficits following α-synuclein PFFs-induced toxicity. Taken together, these findings indicate that Radotinib HCl has beneficial neuroprotective effects in PD and provides strong evidence that selective and brain permeable c-Abl inhibitors can be potential therapeutic agents for the treatment of PD.

These data are very compelling to evaluate the effects of Radotinib in a phase II, randomized, double-blind, placebo-controlled trial in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female from 40 to 80 years old;
2. Diagnosed with "Clinically Probable Parkinson's Disease" according to the MDS clinical diagnostic criteria, with documented onset of symptoms per treating physician's records within three years of the screening visit;
3. Positive DAT-scan (e.g. a striatal dopamine transporter deficit on dopamine transporter imaging by DaT-SPECT, characterized by crescent-shaped areas of asymmetrical aspect, or of symmetrical aspect but of uneven intensity, between the right and the left brain hemisphere) confirmed by local reading;
4. Hoehn & Yahr stage ≤ 2.5;
5. Without previous symptomatic treatment for PD disease and with current clinical state not requiring started dopaminergic therapy within 6 months from Baseline;
6. Absence of a parkinsonian syndrome and other neurovascular comorbidities, confirmed by MRI
7. Female subjects must be not of childbearing potential, e.g., documented evidence that they are surgically sterile (e.g., hysterectomy, partial hysterectomy, bilateral oophorectomy, bilateral tubal ligation), or postmenopausal (at least 12 months since last menses) or using highly effective method of birth control defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as combined hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intra uterine devices (IUDs), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, condom, until at least one month after the last drug intake associated to a negative pregnancy test at screening;
8. Covered by Health Insurance System;
9. Able to understand and to sign the informed consent prior to screening;
10. Blood Pressure (BP) and Heart Rate (HR) considered NCS by Investigator;
11. Electrocardiogram (ECG) recording on a 12-lead ECG considered NCS by Investigator;
12. Laboratory parameters within the normal range of the laboratory. Individual values out of the normal range can be accepted if judged clinically non relevant by the Investigator.

Exclusion Criteria:

1. Atypical Parkinsonism or drug-induced Parkinsonism;
2. Current, or within 60 days of screening, use of any prescription, investigational, or over the counter medication for the symptomatic treatment of PD or to slow the progression of PD.
3. Prior use of dopaminergic therapy (e.g., levodopa, dopamine agonist, amantadine, rasagiline) for 30 or more days any time in the past;
4. Cognitive impairment (MMSE ≤ 24);
5. Active psychiatric disorder (mood disorders, hallucinations or delirium with strong functional impact and not controlled by medication or which happened during the last 3 months before inclusion);
6. Severe or uncontrolled chronic disease;
7. Significant medical history of congenital or acquired bleeding disorders;
8. Treatment by Deep Brain Stimulation or continuous infusion of apomorphin/dopa gel;
9. Any below impaired cardiac function:

   * LVEF <45% or < lower bound of normal limit of study site (whichever higher), confirmed by echocardiogram (if the subject has already carried out this examination during the last month before inclusion, he/she will be exempted from retaking this examination, but he/she will have to present the echocardiogram as well as the cardiologist's report. If not, this exam should be performed during the screening period)
   * Subjects who cannot have QT intervals measured according to ECG
   * Complete left bundle branch block
   * Subjects with cardiac pacemakers
   * Subjects with congenital long QT syndrome or the family history of known long QT syndrome
   * History of, or presence of symptomatic ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia (< 50 bpm).
   * Mean QTcF >450msec following three consecutive ECG tests at baseline: Screening test will be performed again for QTcF after the adjustment of electrolyte if QTcF >450msec and the electrolyte is not within the normal range
   * Medical history of clinically confirmed myocardial infarction
   * Medical history of unstable angina (within last 12 months)
   * Other clinically significant cardiac disease (e.g. congestive heart failure, or uncontrolled hypertension)
10. Participation in other investigational drug trials within 30 days prior to Screening;
11. Any concomitant medication or medication excluded that could put subject at risk, or interfere with study evaluations;
12. Subjects currently receiving treatment with a strong CYP3A4 inhibitors (e.g. erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil) or strong CYP3A4 inducers (e.g. dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbitol, St. John's Wort) or therapeutic Cumarin derivatives (e.g. warfarin, acenocoumarol, phenprocoumon) and that can neither stop the administration of these drugs before the start of the IP administration nor switch to other drugs
13. Subjects who are currently receiving treatment with a medication that has the potential to extend QT intervals and can neither stop the administration of the drugs before the start of the IP administration nor switch to other drugs (list of medications that have the potential to prolong QT interval is provided in the Appendix II) If subjects need to start such drug treatments during the study, this will be discussed with the sponsor, IL-YANG PHARM. Co., Ltd.
14. Subjects who are currently receiving treatment with P-gp inducers (e.g. (Ritonavir, Saquinavir, Nelfinavir, Indinavir, Amprenavir, Tipranavir…), Apalutamide, Estrone, Estriol, Trazodone, Vincristine, Tamoxifen, Doxorubicin, Carbamazepine, Oxcarbazepine, Fosphenytoin, Lorlatinib, Phenobarbital, Phenytoin, Propofol, beclomethasone, Dexamethasone, Prednisone, Hydrocortisone, Diclofenac, Rifampicin, Reserpine, Nifedipine, Digoxine, Amiodarone, Spironolactone, Levothyroxine, Tacrolimus, Sirolimus, St. John's Wort (herbal ingredient)) and that can neither stop the administration of these drugs before the start of the IP administration nor switch to other drugs;
15. Gastrointestinal disorder or gastrointestinal disease that may result in a significant change in the absorption of the investigational product;
16. Medical history of acute or chronic pancreatitis within the past one year;
17. Acute or chronic liver, pancreas, or severe kidney disease that are not associated with the disease;
18. Subjects known seropositive to human immunodeficiency virus (HIV), current acute or chronic hepatitis B (hepatitis B surface-antigen positive), hepatitis C, or cirrhosis. Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA < 500 IU/mL or site specific local lab normal range lower limit assessed by investigator), and cured hepatitis C subjects can be enrolled;
19. Men subjects who are unwilling to use and appropriate method of contraception during the study;
20. Subjects who have hypersensitivity to active ingredient or any of the excipients of this investigational product;
21. Any medical condition that might interfere with the protocol except those defined in Section 5.3 of the study protocol;
22. Subject unable to attend scheduled visits or to comply to the protocol;
23. Subject under legal guardianship or judicial protection;
24. Subject in the exclusion period of another protocol;
25. No possibility of contact in case of emergency.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety parameters: Adverse Events | 12 months after dose administration
  Incidence and severity of treatment emergent AEs

SECONDARY OUTCOMES:
Pharmacokinetics assessments of Radotinib HCl: Cmax | 14 days after dose administration
  The maximum (peak) observed drug concentration after dose administration
Pharmacokinetics assessments of Radotinib HCl: Tmax | 14 days after dose administration
  The time to reach maximum (peak) drug concentration after dose administration
Pharmacokinetics assessments of Radotinib HCl: Ctrough | 14 days after dose administration
  Trough plasma concentration (measured concentration at the end of a dosing interval at steady state)
Pharmacokinetics assessments of Radotinib HCl: AUCt | 14 days after dose administration
  Area under the plasma concentration-time curve from time zero to time t
Pharmacokinetics assessments of Radotinib HCl: AUCinf | 14 days after dose administration
  Area under plasma concentration-time curve from time 0 to infinity
Pharmacokinetics assessments of Radotinib HCl: AUC0-12h | 14 days after dose administration
  Area under the plasma concentration-time curve over the last 24-h dosing interval
Pharmacokinetics assessments of Radotinib HCl: t1/2 | 14 days after dose administration
  Elimination half-life of Radotinib after dose administration
Pharmacokinetics assessments of Radotinib HCl: Vd/F | 14 days after dose administration
  Apparent volume of distribution after non-intravenous administration
Pharmacokinetics assessments of Radotinib HCl: CL/F | 14 days after dose administration
  Apparent total clearance of the drug from plasma after oral administration
Change from Baseline in the sum of MDS-UPDRS Parts I, II and III | 6 months
  The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is a clinimetric assessment of subjective and objective symptoms and signs of Parkinson's disease created by the Movement Disorder Society.
  The MDS-UPDRS has four parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living, Part III (motor examination) and Part IV (motor complications). Only Parts I, II and III will be completed in this study.
  MDS-UPDRS retains the four-scale structure with a reorganization of the various subscales. The subscale has a 0-4 rating, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. Higher MDS-UPDRS scores reflect worse tremor/motor function. Larger differences will infer greater effect size for the intervention. Score drops over time imply improvement in tremor/motor function.
Time from baseline to initiation of dopamine-replacement medication. | 6 months
  Time from baseline to initiation of dopamine replacement therapy following randomization
Change in health related quality of life as measured by a quality of life questionnaire (PDQ-39) | 12 months
  The Parkinson's Disease Questionnaire (PDQ-39) is a 39-item quality of life questionnaire for patients with Parkinson's Disease (PD) that evaluates the 8 dimensions of mobility, activities of daily living, emotional well-being, stigma, social support, cognition, and communication. The PDQ-39 Single Index (SI) score is the weighted addition of scores on all 8 dimension and ranges from 0 (no disease impact) to 100 (severe disease impact).
Subject's clinical global impression of change. | 12 months
  The CGI Scale of Global Clinical Impressions (see Appendix VI) allows an overall assessment of the subject's condition. The CGI addresses the majority of mental disorders. In its first item, rated from 1 to 7 (the rating 1 corresponding to the normal state), it allows a good overall measurement of the subject's condition. The 2nd item proposes to the Investigator to evaluate the overall improvement of the subject compared to his/her condition at the admission to the research. As before, this item has 7 quantified degrees (from 1 = "very strongly improved" to 7 = "very strongly aggravated").

OTHER OUTCOMES:
Brain DaT SPECT to measure dopamine neurons and nerve terminals | 12 months
  DaTscan is a specific type of single-photon emission computed tomography (SPECT) imaging technique that helps visualize dopamine transporter in the brain
Concentration of α-synuclein in CSF | 6 months
  Quantification of α-synuclein concentration in CSF
Concentration of Tau and phospho-Tau (p-181) in CSF | 6 months
  Quantification of Tau and phospho-Tau (p-181) concentration in CSF
Concentration of β-amyloid peptide 1-42 in CSF | 6 months
  Quantification of β-amyloid peptide 1-42 concentration in CSF
Concentration of NF-L in the serum | 6 months
  Quantification of NF-L concentration in CSF
Concentration of Radotinib HCl in the CSF and plasma | 6 months
  Quantification of Radotinib HCl concentration in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DAMIER, Pr., Principal Investigator — CHU Nantes - Hôpital Nord Guillaume et René Laennec
Locations (7):
- France (7):
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - CHU Limoges, Limoges
  - CHU de Lyon HCL, Lyon
  - Hôpital Nantes-Hotel Dieu, Nantes
  - Hôpital Pitié-Salpêtrière, Paris
  - Chu La Miletrie, Poitiers
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102